CLINICAL TRIAL: NCT07083908
Title: Sphincter Pressures in Women With Obstetric Anal Sphincter Injury: A Comparison of THD® Anopress With High Resolution Anorectal Manometry
Brief Title: A Comparison of THD® Anopress With High Resolution Anorectal Manometry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 350163
Record Dates: First submitted 2025-02-26; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-11

CONDITIONS: Obstetric Anal Sphincter Injury

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- THD® Anopress (Sensyprobe) first (Other)
  Interventions: Device: THD® Anopress (Sensyprobe) first
- High Resolution Anorectal Manometry first (Other)
  Interventions: Device: High Resolution Anorectal Manometry first

INTERVENTIONS:
Device: THD® Anopress (Sensyprobe) first — Anorectal manometry with THD® Anopress (Sensyprobe) first then with High Resolution Anorectal Manometry (Laborie)
  Arms: THD® Anopress (Sensyprobe) first
Device: High Resolution Anorectal Manometry first — Anorectal manometry with High Resolution Anorectal Manometry (Laborie) first followed by THD® Anopress (Sensyprobe)
  Arms: High Resolution Anorectal Manometry first

SUMMARY:
Currently, high resolution anorectal manometry (HDARM) is used as gold standard to measure anal sphincter pressures in women who have sustained a third or fourth degree perineal tears (obstetric anal sphincter injuries). This test is performed to help advise patients on future pregnancies or deliveries. However, HDRM catheters are very expensive and they also need to be performed in a dedicated procedure room. THD® Anopress in comparison is a lightweight, portable device which has a comparatively shorter investigation time and is more cost- effective.

However, although THD® Anopress is currently used in the colorectal population, there is currently no validated research that compares the measurements obtained by HDARM with that of THD® Anopress with women with a history of obstetric anal sphincter injuries.

The primary aim of this study is to compare pressure measurements from HDARM to that of THD® Anopress in women with obstetric anal sphincter injuries.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with a history of obstetric anal sphincter injury and are:

   a) At least 6 weeks postpartum
2. Either able to speak, read and write in English, or has a professional interpreter present at the time of appointment.
3. Capable of understanding and signing the informed consent form after full discussion of the investigations and its risks and benefits.
4. Able and willing to complete the St Mark's Score, ICIQ-UI SF and other trial related questionnaires, comply with scheduled clinic visits and manometry studies.

Exclusion Criteria:

1. Existing anal pain precluding anorectal examination
2. Neurological conditions such as stroke, multiple sclerosis, spinal cord injury or Parkinson's disease
3. Age <18 years old
4. Currently pregnant -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Main voluntary squeeze increment | Day 1
  Difference between maximum voluntary squeeze pressure and maximum resting pressure (mmHg)

SECONDARY OUTCOMES:
Anal resting pressure (mmHg) | Day 1
  Agreement/ accuracy of manometric values of THD® Anopress compared with HD-ARM on anal resting pressures (mmHg)
Main voluntary squeeze increment | Day 1
  difference between maximum voluntary squeeze pressure and maximum resting pressure (mmHg)
Endurance squeeze pressure | Day 1
  Agreement/ accuracy of manometric values of THD® Anopress compared with HD-ARM on endurance squeeze pressures (increase of average pressure within 5 seconds of maximum squeeze) (mmHg)
Straining pressure | Day 1
  Agreement/ accuracy of manometric values of THD® Anopress compared with HD-ARM on straining pressure (mmHg)
Total duration of procedure | Day 1
  Time from commencement to end of procedure (minutes and seconds)
Visual Analogue Scale (VAS) | Day 1
  Visual Analogue Scale -10 points (0-10), with 0 being 'no pain' and 10 being 'worst pain imaginable'
Adverse events | Day 1
  Any adverse reactions ie. patient injury, severe discomfort, medical emergencies encountered

CONTACTS AND LOCATIONS:
Locations (1):
- Kings College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No